CLINICAL TRIAL: NCT00251420
Title: Writing About Disease: Effect on Rehabilitation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LHL Helse (Other)
Collaborators: The norwegian association for heart and lung patients (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: G22-1
Record Dates: First submitted 2005-11-09; First posted 2005-11-10 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: COPD; Asthma
Keywords: copd; asthma; QoL; Perceived health status; Trait anxiety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: writing about disease — writing about physical or emotional consequences of pulmonary disease

SUMMARY:
Therapeutic writing about one's emotions has been described previously (J Pennebaker: Emotions, disclosure and health. Am Psychol. Assoc 1995). The present project will compare the effects (if any) of writing about the emotional versus the physical consequences of lung disease on anxiety, perceived quality of life, and perceived health status.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) patients (age 35-70) and asthma patients (age 20-60) referred to a 4 weeks inpatient rehabilitation program - who agree to participate in the project - are randomly assigned to one of three conditions:

* Writing about emotional consequences of their disease before the program starts
* Writing about physical consequences of their disease before the program starts
* Not writing

All patients are measured (completing questionnaires at home) on: perceived quality of life, perceived health status and trait anxiety - 2 weeks before the program, 2 weeks after the program and 6 months after the program. FEV1 and 6 min walking distance are measured at the beginning and by the end of the program.

In addition to questionnaires, all patients are asked to:

* Write in their own words ( 2 weeks after) to evaluate their stay at the rehabilitation clinic; and
* Write in their own words (6 months after) about how the disease affects their life at that point.

Both quantitative and qualitative data will be used for analysis purposes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD (age between 35 and 70)
* Clinical diagnosis of asthma (age between 20 and 60)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-12; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Quality of life | prospective
Perceived health status | prospective
Trait anxiety | prospective

SECONDARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | prospective
6-minute walking distance | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Einar Haave, Cand Psychol, Principal Investigator — LHL Helse
Locations (1):
- Glittreklinikken, Hakadal, Akershus, Norway